CLINICAL TRIAL: NCT03809468
Title: Patient Satisfaction With Initial Phone Call Versus Office Visit Following Minimally Invasive Hysterectomy, a Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FLA 18-095
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Abnormal Uterine Bleeding
Keywords: patient satisfaction, hysterectomy, follow up
MeSH Terms: conditions — Metrorrhagia; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Routine follow up of a clinic visit at 1-2 weeks postop, and 6-8 weeks postop.
- study (Experimental): phone call follow up instead of clinic visit follow up at 1-2 weeks, followed by 6-8 week clinic follow up
  Interventions: Other: phone call follow up

INTERVENTIONS:
Other: phone call follow up — instead of a clinic visit, patients will be randomized to a phone call
  Arms: study

SUMMARY:
Patients will be randomized to clinic or telephone follow up after outpatient TLH. surveys will document patient satisfaction.

DETAILED DESCRIPTION:
This is a randomized controlled trial looking at patient satisfaction with a 1-2 week postoperative visit versus phone call after minimally invasive hysterectomy. Patients will be screened, enrolled, consented, and randomized during the preoperative office encounter, which usually takes place 30 days prior to their scheduled surgery. Patients randomized to the study group (1-2 week postoperative phone call) will be given a time and date when to expect the postoperative phone call. Patients randomized to the control arm will receive a standard postoperative visit appointment 7-21 days after surgery. Patients in both arms will receive postoperative discharge instructions advising when to contact our office and when to present to the emergency room with certain complaints. The patients in the study arm will have instructions reinforcing that they will be contacted with a postoperative phone call instead of a visit initially; however, patients in both arms will have a postoperative visit 6-8 weeks following surgery.

After surgery, patients randomized to the study arm will receive the phone call at 7-14 days post-op. The physician performing the phone call will be a minimally invasive gynecology fellow in our practice. The provider will use a script to review all of the typical review of systems and pertinent postoperative functioning questions typically reviewed and documented in our postoperative visit. They will also review the surgical pathology at this time. This conversation will be documented in our electronic medical record.

Patients randomized to the control arm will undergo typical office visit at 7-21 days postop.

Patients in both arms will have postoperative office visits at 6-8 weeks postop, and will complete a survey at that time. The survey is a modified version of the SCAHPS survey to assess patient satisfaction with the surgical experience. There will also be some questions about the patients' attitudes towards the number and timing of postoperative visits.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing minimally invasive hysterectomy

Exclusion Criteria:

* patients without adequate phone or transportation access
* patients with concern for underlying malignancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 6-8 weeks postop
  patient satisfaction scores

SECONDARY OUTCOMES:
phone calls and visits (unplanned) | 6-8 weeks postop

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Frazzini Padilla, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States